CLINICAL TRIAL: NCT05713903
Title: Comparison of Laparoscopic Versus Open Right Colectomy for Right Colon Cancer, According to the Complete Mesocolic Excision (CME) Principles: a Prospective Randomized Controlled Trial
Brief Title: Laparoscopic Versus Open Right Colectomy for Right Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Perivoliotis Konstantinos, Perivoliotis Konstantinos, Principal Investigator, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LORC
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer
Keywords: colon; cancer; open; laparoscopic; colectomy; right; mesocolic; excision
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective, parallel randomized-controlled design
Masking Description: There will be no blindness at the level of the patient, the treating physicians (surgeon, anesthesiologist) and the researcher who will record the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic right colectomy (Experimental): In laparoscopic right colectomy subgroup, the patient will be placed in a lithotomy position. Entrance in the peritoneal cavity will be completed via the open Hasson method. Overall, 4 ports will be used: 10mm at the umbilicus for optical entry, 12mm in the left midclavicular line below the umbilicus as the main working port, 5mm at the McBurney point, and 5mm between the umbilicus and the xiphoid process. Dissection of the peritoneal fold, under the terminal ileum, will be performed based on the medial to lateral approach. Similar to the open approach, the ileocolic vessels, as well as the right branches of the middle colic will be ligated at their origin for cecal and proximal ascending tumors. For hepatic flexure cancers, the medial colic vessels will be ligated. The ileocolic anastomosis will be completed either intracorporeally or extracorporeally, using staples or sutures.
  Interventions: Procedure: Laparoscopic right colectomy
- Open right colectomy (Active Comparator): In the open right colectomy group, the operation will start with a midline incision and dissection based on the lateral to medial approach. The lateral peritoneal fold along Toldt's line will be incised and the ascending colon will be mobilized from the retroperitoneum according to the embryological dissection planes. Dissection will continue until the anterior surface of the superior mesenteric vessels at the third duodenal part. Ileocolic and right colic vessels will be ligated at their origins. For hepatic flexure tumors, the middle colic vessels will be also ligated at their origin. The ileocolic anastomosis will be performed using an automatic stapler. The anastomosis will be completed either with staples or sutures.
  Interventions: Procedure: Open right colectomy

INTERVENTIONS:
Procedure: Laparoscopic right colectomy — Resection of the ascending colon via a laparoscopic approach, adhering to the CME principles
  Arms: Laparoscopic right colectomy
Procedure: Open right colectomy — Resection of the ascending colon via an open approach, adhering to the CME principles
  Arms: Open right colectomy

SUMMARY:
The purpose of this research protocol is to compare open versus laparoscopic right colectomy (according to the CME technique of complete mesocolic excision) for right colon cancer. This study will be designed as a prospective randomized controlled trial. The comparison of the two techniques will include endpoints regarding the quality characteristics of the specimens and the oncological results. In addition, the effectiveness of the two methods will be evaluated in terms of the early and late postoperative period.

DETAILED DESCRIPTION:
Colorectal cancer is the third and second most common malignancy in male and female patients, respectively, with up to 1.8 million new cases and 860,000 deaths per year.

Anterior resection with total mesorectal excision (TME) was first proposed by Heald in 1982 and is currently the gold standard surgical technique for middle and lower rectal cancer. Heald considered that the metastatic spread of the tumor occurs through micro-implantations in the lymph node network of the mesorectum, and much less through horizontal intramural infiltration, and thus defined rectal resection margins at 5cm or even 2cm for well-differentiated neoplasms. Therefore, he suggested that mesorectum displays a greater risk for micro-metastatic disease and should be removed en-bloc with intact resection margins.

Similarly in 2009, Hohenberger proposed the complete mesocolon excision (CME) concept for the treatment of colon cancer, based on the respective embryological development anatomical planes. After analyzing a large cohort of patients, he concluded that this operation type leads to a significant reduction in the local recurrence and an increase in the overall survival rates.

Hohenberger proposed open CME as the optimal surgical technique for colon cancer, under the premise that the following principles are met:

* Dissection of Toldt's fascia and mesocolon preservation
* Central vascular ligation
* Extensive locoregional lymph node dissection CME technique, as described by Hohenberger in 2008, is an extension of Heald's TME and it is based on the sharp dissection and separation of the visceral fascia that surrounds the colon from the parietal fascia. The aim is to fully mobilize the colon and the corresponding mesocolon, which is surrounded bilaterally by sheets of visceral fascia. This ensures the complete resection of the tumor and the corresponding lymph nodes. At the same time, central vascular ligation allows the dissection of the apical lymph nodes.

There are three resection planes: the mesocolic, intramesocolic and muscularis propria plane. The ideal resection plane is the mesocolic, in which the colon is removed, along with the entire mesocolon and all the venous and lymphatic tissue, without violating the visceral fascia. Surgical specimens categorized into either of the other two resection planes are associated with reduced R0 resection rates and with reduced overall survival. Characteristically, the muscularis propria resection plane has been associated with up to 15% reduced survival rate compared to the mesocolic plane.

There are specific morphometric characteristics of surgical specimens that are used to assess their quality. These include tumor and proximal colon high vascular ligation distance, number of lymph nodes, length of resected small bowel and colon, and total area of the mesocolon. These characteristics are directly related to the number of harvested lymph nodes and, therefore, to overall survival.

According to initial results, CME specimens were larger in size, contained a longer length of colon, a larger mesenteric surface and a greater number of lymph nodes compared to the standard colectomy specimens. In addition, a greater distance of the tumor from the resection margins was highlighted. Specifically for right colon cancers, recent publications have shown that CME can achieve better morphometric specimen characteristics and a greater number of lymph nodes. In a recent randomized study, Di Buono et al. compared the completion of CME or not, during laparoscopic right colectomy. A significant difference was found in favor of CME, regarding the specimen length and the lymph node harvest.

Despite these, the literature evidence regarding the morphological and qualitative characteristics of laparoscopic and open CME specimens are still inconclusive. Specifically for right colectomies, in the comparative study by Gouvas et al., it was observed that the percentage of the mesocolic resection level was 100% in open colectomy, in contrast to 85.7% in the laparoscopic approach. However, this difference was not statistically significant. In a retrospective study by Ali Koc et al., no difference was found between open and laparoscopic CME in terms of specimen length, R0 resection rate and number of resected lymph nodes. A recent publication by Ali Zedan et al., argued that open CME is associated with longer specimens, larger mesenteric area, and increased resection margins. Another interesting finding was that the number of lymph nodes and the distance of the ligation site were greater in the laparoscopic CME group. However, the meta-analysis by Anania et al. failed to validate any difference between the two methods in the total number of lymph nodes. Finally, a comparative analysis of our own series of patients did not show superiority of one technique over the other in terms of resection level, specimen length and number of lymph nodes.

Additional qualitative characteristics of a colon cancer operation include operative time, intraoperative blood loss, time of bowel function recovery, length of postoperative hospital stay, postoperative complications, as well as overall survival and local recurrence rate. In a recent meta-analysis by Anania et al. applying the principles of CME to right colectomies did not affect the rates of postoperative leaks, bleeding, overall complications, and reoperations. However, CME right colectomy was associated with optimal results in terms of 3-year overall survival and 5-year disease-free survival.

Regarding the application of laparoscopy principles to CME colectomies, previous studies have confirmed that it is a technique with optimal results, such as faster postoperative recovery, shorter hospital stay, and lower morbidity. There is agreement between studies regarding the perioperative benefits of laparoscopic CME right colectomy versus the open method. According to Huang et al., the length of operative time between the two techniques was comparable. Laparoscopic right colectomy was associated with significantly lower intraoperative blood loss and faster initiation of feeding. In addition, these patients were discharged earlier compared to their counterparts in the open colectomy group. Moreover, no differences were observed in complication and local recurrence rates. These findings were also confirmed by the comparative study of Sheng et al., where the application of the minimally invasive technique resulted in lower levels of postoperative pain, and faster recovery. Accordingly, Shin et al., applying propensity score analysis, to remove possible confounding factors, in a sample of 2249 right colectomies and found that the technique is an independent predictor for 5-year disease-free survival. Pooled data from Anania et al., confirmed the superiority of laparoscopic CME in the rates of postoperative complications, intraoperative bleeding, and length of hospital stay. These are also in accordance with our own experience, where a significant benefit of the laparoscopic approach was shown in the duration of hospitalization and septic complications, at the cost of prolonged surgical time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed right colon cancer (cecum, ascending colon, hepatic flexure)
* Surgical resection based on the CME principles
* Patient 18 to 90 years old
* American Society of Anesthesiologists score ≤III
* Τ≤3
* Elective operation
* Signed informed consent of the patient

Exclusion Criteria:

* Non elective operation (hemorrhage, perforation, obstruction)
* Locally advanced disease (T4)
* Distant metastases (Stage IV)
* American Society of Anesthesiologists ≥IV
* Previous laparotomy
* BMI >35 kg/m2
* Active sepsis or systemic infection
* Untreated physical and mental disability
* Pregnancy or breast-feeding
* Lack of compliance with the protocol process
* Non-granting of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Mesocolic Resection Plane | 1 month postoperatively
  Occurrence of Mesocolic Resection Plane. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'

SECONDARY OUTCOMES:
Open Conversion | Intraoperative period
  Occurrence of Open Conversion. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Operative Time | Intraoperative period
  The total operative time will be recorded. Measurement unit: minutes
Type of Anastomosis | Intraoperative period
  Occurrence of Stapled or Handsewn Anastomosis. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Intraoperative Transfusion | Intraoperative period
  Occurrence of Intraoperative Transfusion. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Postoperative Complication | 1 month postoperatively
  Occurrence of Postoperative Complication. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Bowel Function Recovery | 7 days postoperatively
  Postoperative time until the recovery of bowel function is achieved. Measurement unit: days
Length of Hospital Stay | Maximum time frame 39 days postoperatively]
  Postoperative time that the patient can be safely discharged. Measurement unit: days. The patient will be discharged, when it is ensured that is medically safe to be released. In particular, as the exit time of the patient, will be regarded the time that the patient will fulfil the Clinical Discharge Criteria
Negative Resection Margin | 1 month postoperatively
  Occurrence of Negative Resection Margin. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Local Recurrence | 5 years postoperatively
  Occurrence of Local Recurrence. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Disease Free Survival | 5 years postoperatively
  Occurrence of Disease Free Survival. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'
Overall Survival | 5 years postoperatively
  Occurrence of Overall Survival. If such an episode occurs, then it will be defined as=1 'YES' If such an episode does not occur, then it will be defined as=0 'NO'

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Perivoliotis, MD, Principal Investigator — University Hospital of Larissa; George Tzovaras, Prof, Study Chair — University Hospital of Larissa; Ioannis Baloyiannis, Prof, Study Director — University Hospital of Larissa
Locations (1):
- Department of Surgery, University Hospital of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data

REFERENCES:
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Hohenberger W, Weber K, Matzel K, Papadopoulos T, Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation--technical notes and outcome. Colorectal Dis. 2009 May;11(4):354-64; discussion 364-5. doi: 10.1111/j.1463-1318.2008.01735.x. Epub 2009 Nov 5. PMID 19016817
- [Background] Strey CW, Wullstein C, Adamina M, Agha A, Aselmann H, Becker T, Grutzmann R, Kneist W, Maak M, Mann B, Moesta KT, Runkel N, Schafmayer C, Turler A, Wedel T, Benz S. Laparoscopic right hemicolectomy with CME: standardization using the "critical view" concept. Surg Endosc. 2018 Dec;32(12):5021-5030. doi: 10.1007/s00464-018-6267-0. Epub 2018 Oct 15. PMID 30324463
- [Background] Matsuda T, Iwasaki T, Sumi Y, Yamashita K, Hasegawa H, Yamamoto M, Matsuda Y, Kanaji S, Oshikiri T, Nakamura T, Suzuki S, Kakeji Y. Laparoscopic complete mesocolic excision for right-sided colon cancer using a cranial approach: anatomical and embryological consideration. Int J Colorectal Dis. 2017 Jan;32(1):139-141. doi: 10.1007/s00384-016-2673-8. Epub 2016 Oct 6. PMID 27714518
- [Background] Gouvas N, Pechlivanides G, Zervakis N, Kafousi M, Xynos E. Complete mesocolic excision in colon cancer surgery: a comparison between open and laparoscopic approach. Colorectal Dis. 2012 Nov;14(11):1357-64. doi: 10.1111/j.1463-1318.2012.03019.x. PMID 22390358
- [Background] West NP, Hohenberger W, Weber K, Perrakis A, Finan PJ, Quirke P. Complete mesocolic excision with central vascular ligation produces an oncologically superior specimen compared with standard surgery for carcinoma of the colon. J Clin Oncol. 2010 Jan 10;28(2):272-8. doi: 10.1200/JCO.2009.24.1448. Epub 2009 Nov 30. PMID 19949013
- [Background] Siani LM, Lucchi A, Berti P, Garulli G. Laparoscopic complete mesocolic excision with central vascular ligation in 600 right total mesocolectomies: Safety, prognostic factors and oncologic outcome. Am J Surg. 2017 Aug;214(2):222-227. doi: 10.1016/j.amjsurg.2016.10.005. Epub 2016 Nov 16. PMID 27876380
- [Background] Hurwitz EE, Simon M, Vinta SR, Zehm CF, Shabot SM, Minhajuddin A, Abouleish AE. Adding Examples to the ASA-Physical Status Classification Improves Correct Assignment to Patients. Anesthesiology. 2017 Apr;126(4):614-622. doi: 10.1097/ALN.0000000000001541. PMID 28212203
- [Background] Wang Y, Zhang C, Zhang D, Fu Z, Sun Y. Clinical outcome of laparoscopic complete mesocolic excision in the treatment of right colon cancer. World J Surg Oncol. 2017 Sep 18;15(1):174. doi: 10.1186/s12957-017-1236-y. PMID 28923055
- [Background] Feng B, Sun J, Ling TL, Lu AG, Wang ML, Chen XY, Ma JJ, Li JW, Zang L, Han DP, Zheng MH. Laparoscopic complete mesocolic excision (CME) with medial access for right-hemi colon cancer: feasibility and technical strategies. Surg Endosc. 2012 Dec;26(12):3669-75. doi: 10.1007/s00464-012-2435-9. Epub 2012 Jun 26. PMID 22733200
- [Background] Adamina M, Manwaring ML, Park KJ, Delaney CP. Laparoscopic complete mesocolic excision for right colon cancer. Surg Endosc. 2012 Oct;26(10):2976-80. doi: 10.1007/s00464-012-2294-4. Epub 2012 May 2. PMID 22549374
- [Background] Kang J, Kim IK, Kang SI, Sohn SK, Lee KY. Laparoscopic right hemicolectomy with complete mesocolic excision. Surg Endosc. 2014 Sep;28(9):2747-51. doi: 10.1007/s00464-014-3521-y. Epub 2014 Apr 10. PMID 24718666
- [Background] Di Buono G, Buscemi S, Cocorullo G, Sorce V, Amato G, Bonventre G, Maienza E, Galia M, Gulotta L, Romano G, Agrusa A. Feasibility and Safety of Laparoscopic Complete Mesocolic Excision (CME) for Right-sided Colon Cancer: Short-term Outcomes. A Randomized Clinical Study. Ann Surg. 2021 Jul 1;274(1):57-62. doi: 10.1097/SLA.0000000000004557. PMID 33177355
- [Background] Anania G, Davies RJ, Bagolini F, Vettoretto N, Randolph J, Cirocchi R, Donini A. Right hemicolectomy with complete mesocolic excision is safe, leads to an increased lymph node yield and to increased survival: results of a systematic review and meta-analysis. Tech Coloproctol. 2021 Oct;25(10):1099-1113. doi: 10.1007/s10151-021-02471-2. Epub 2021 Jun 12. PMID 34120270
- [Background] Koc MA, Celik SU, Guner V, Akyol C. Laparoscopic vs open complete mesocolic excision with central vascular ligation for right-sided colon cancer. Medicine (Baltimore). 2021 Feb 12;100(6):e24613. doi: 10.1097/MD.0000000000024613. PMID 33578570
- [Background] Zedan A, Elshiekh E, Omar MI, Raafat M, Khallaf SM, Atta H, Hussien MT. Laparoscopic versus Open Complete Mesocolic Excision for Right Colon Cancer. Int J Surg Oncol. 2021 Feb 2;2021:8859879. doi: 10.1155/2021/8859879. eCollection 2021. PMID 33604087
- [Background] Anania G, Arezzo A, Davies RJ, Marchetti F, Zhang S, Di Saverio S, Cirocchi R, Donini A. A global systematic review and meta-analysis on laparoscopic vs open right hemicolectomy with complete mesocolic excision. Int J Colorectal Dis. 2021 Aug;36(8):1609-1620. doi: 10.1007/s00384-021-03891-0. Epub 2021 Mar 1. PMID 33644837
- [Background] Magouliotis DE, Baloyiannis I, Mamaloudis I, Bompou E, Papacharalampous C, Tzovaras GA. Laparoscopic Versus Open Right Colectomy for Cancer in the Era of Complete Mesocolic Excision with Central Vascular Ligation: Pathology and Short-Term Outcomes. J Laparoendosc Adv Surg Tech A. 2021 Nov;31(11):1303-1308. doi: 10.1089/lap.2020.0508. Epub 2021 Mar 12. PMID 33719562
- [Background] Huang JL, Wei HB, Fang JF, Zheng ZH, Chen TF, Wei B, Huang Y, Liu JP. Comparison of laparoscopic versus open complete mesocolic excision for right colon cancer. Int J Surg. 2015 Nov;23(Pt A):12-7. doi: 10.1016/j.ijsu.2015.08.037. Epub 2015 Aug 28. PMID 26318966
- [Background] Sheng QS, Pan Z, Chai J, Cheng XB, Liu FL, Wang JH, Chen WB, Lin JJ. Complete mesocolic excision in right hemicolectomy: comparison between hand-assisted laparoscopic and open approaches. Ann Surg Treat Res. 2017 Feb;92(2):90-96. doi: 10.4174/astr.2017.92.2.90. Epub 2017 Jan 31. PMID 28203556
- [Background] Shin JK, Kim HC, Lee WY, Yun SH, Cho YB, Huh JW, Park YA, Chun HK. Laparoscopic modified mesocolic excision with central vascular ligation in right-sided colon cancer shows better short- and long-term outcomes compared with the open approach in propensity score analysis. Surg Endosc. 2018 Jun;32(6):2721-2731. doi: 10.1007/s00464-017-5970-6. Epub 2017 Nov 3. PMID 29101572
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05713903/Prot_002.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05713903/ICF_003.pdf